CLINICAL TRIAL: NCT02859012
Title: Randomized Phase II Study of Axitinib in Patients With Recurred or Metastatic Adenoid Cystic Carcinoma
Brief Title: Study of Axitinib in Patients With Recurred or Metastatic Adenoid Cystic Carcinoma
Acronym: AxitinibACC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Bhumsuk Keam, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Axitinib in ACC
Record Dates: First submitted 2016-07-28; First posted 2016-08-08 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Recurrent ACC, metastaticACC, Unreaectable ACC
MeSH Terms: interventions — Axitinib; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- axitinib (Experimental): Axitinib 5 mg twice (10mg) daily po medication until progression or development of unacceptable toxicity (4 weeks is considered as one cycle).
  Interventions: Drug: Axitinib
- observation (Active Comparator): Observation. if disease progression is detected, cross-over will be permitted.
  Interventions: Other: Observation

INTERVENTIONS:
Drug: Axitinib — Dosing schedule: 5mg twice per day orally (4 weeks is considered as 1 cycle)
  Other Names: Inlyta
  Arms: axitinib
Other: Observation — this group is observational ones.
  Arms: observation

SUMMARY:
To understand efficacy of axitinib in recurred or metastatic adenoid cystic carcinoma

DETAILED DESCRIPTION:
Adenoid cystic carcinoma (ACC) is a rare variant of adenocarcinoma that occurs in secretory glands such as in salivary glands. Although ACC is histologically low grade and slow-growing, more than half of patients eventually have recurrent and/or metastatic disease.

The natural course of metastatic disease with ACC is relatively indolent; however, most patients with metastatic disease ultimately die from their cancer. The management of recurred / metastatic ACC is a distinct therapeutic challenge because of its insidious local growth pattern, propensity for perineural involvement, tendency for distant metastasis, and pronounced ability to recur over a prolonged period.

2. Current treatment

The role of systemic chemotherapy in ACC is very limited and objective response to any cytotoxic or molecular targeted agent is infrequent, and the optimum regimen is unclear. Because of the rarity of ACC, there are few clinical trials investigating the efficacy of systemic chemotherapy. Recurrent/metastatic ACC is an incurable disease with no standard treatments.

VEGF is highly expressed in ACC and its expression correlates with stage, tumor size, vascular invasion, recurrence and metastasis. High expression of VEGF and Ki-67 were independent poor prognostic factors in ACC. MYB/NFIB translocation has recently identified in ACC and MYB protein over expression was found in ACC. MYB over-expression in ACC has been correlated to the increased expression of genes involved in vascular endothelial growth factor (VEGF), KIT . More than 70% of ACCs highly express the oncogenic transcription factor c-myb, which drives expression of genes that activate VEGFR and c-kit pathways.

Several lines of evidence suggest a function for VEGF, PDGFR signaling in ACC progression. The expressions of NF-kappaB p65, iNOS, and VEGF were related with microvessel density. In vitro, the inhibition of VEGF expression via iNOS gene induced apoptosis of ACC cell lines.

Axitinib (AG-013736; Pfizer) is a multi-targeted small-molecule inhibitor of the receptor tyrosine kinases involved in tumor proliferation and angiogenesis, including VEGFR-1, VEGFR-2 and VEGFR-3, c-kit, platelet-derived growth factor receptor (PDGFR)-α and PFGFR-β. Axitinib (AG-013736) has demonstrated a partial response lasting 4 months in one patient with ACC in a phase I trial . In that aspect, Ho et al. conducted phase II study with axitinib in ACC. Interestingly, response rate was 9.1% and tumor shrinkage was observed in 66.7%

Besides of axitinib, other antiangiogenic agents such as sutene or dovitinib showed promising activity in ACC. Dovitinib, which is pan FGFR , VEGF, PDGFR inhibitor showed one confirmed partial response PR (3.1%) and three unconfirmed PR (9.3%). Interestingly, hyperphosphatemia was not observed in this study, and one PR patients showed strong PDGFR beta positivity, which suggests that antiangiogenic pathway is more important than FGFR pathway.

3. Gap, issue or problem that needs to be addressed

Based on these evidences which suggest a function for VGFR, PDGFR signaling in ACC tumorigenesis and progression, the use of axitinib is reasonable and valuable.

However, the huge gap in ACC trial is lack of randomization trial. Until now, there is no randomized trial in ACC because of its rarity. Hence there is no confirmatory trial in ACC. Without randomization trial, we can not say the real efficacy of axitinib.

So we design multicenter randomized trial of axtinib in ACC to confirm the efficacy of axitinib in this orphan disease.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenoid cystic carcinoma
2. Local, locally-advanced or metastatic disease documented as having shown progression on a scan (CT, MRI, MIBI scan) or X-ray taken >9 months prior to baseline compared to a previous image. Progression must be documented according to RECIST 1.1 criteria.
3. Disease that is not amenable to surgery, radiation or combined modality therapy with curative intent
4. Presence of at least one measurable target lesion for further evaluation according to RECIST 1.1 criteria
5. 18 years or older
6. ECOG performance status 0, 1
7. Adequate organ function

   * ANC ≥ 1500/ μL
   * Platelets ≥100,000/ μL
   * Hemoglobin ≥ 9.0 g/dL
   * Serum creatinine ≤1.5 x ULN
   * Serum bilirubin ≤1.5 x ULN
   * AST, ALT, ≤3.0 x ULN (regardless of liver metastasis)
8. A patient with the willingness to comply with the study protocol during the study period and capable of complying with it
9. A patient who signed the informed consent prior to the participation of the study and who understands that he/she has a right to withdrawal from participation in the study at any time without any disadvantages.

Exclusion Criteria:

1. A patient with no measurable disease
2. Prior chemotherapy, radiation therapy or surgery within 4 weeks prior to study entry except palliative radiotherapy to non-target lesions (within 2 weeks prior to study entry)
3. A patient with intestinal obstruction or impending obstruction, recent active upper GI bleeding
4. A pregnant or lactating patient
5. A patient of childbearing potential without being tested for pregnancy at baseline or with being tested for positive. (A postmenopausal woman with the amenorrhea period of at least 12 months or longer is considered to have non-childbearing potential)
6. A man or woman of childbearing potential who has no willingness to use a contraceptive measure during the study
7. A patient with history of another malignant disease within past 5 years, except curatively treated basal cell carcinoma of skin, early gastric cancer and cervical carcinoma in situ.
8. A patient with history of uncontrolled seizures, central nervous system disorder or psychiatric disorders that are considered clinically significant by the investigator that would prohibit the understanding of informed consent or that may be considered to interfere with the compliance of the administration of the study medications.
9. A patient with clinically significant heart disease (e.g. congestive heart failure, symptomatic coronary artery diseases, cardiac arrhythmia, etc) or myocardial infarction within past 12 months.
10. A patient with organ transplantation requiring immunosuppressive therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate | 6 months

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 year
response rate | 1 year
overall survival | 1 year
duration of response | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bhumsuk Kim, Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Department of Internal Medicine, Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kang EJ, Ahn MJ, Ock CY, Lee KW, Kwon JH, Yang Y, Choi YH, Kim MK, Ji JH, Yun T, Nam BH, Kim SB, Keam B. Randomized Phase II Study of Axitinib versus Observation in Patients with Recurred or Metastatic Adenoid Cystic Carcinoma. Clin Cancer Res. 2021 Oct 1;27(19):5272-5279. doi: 10.1158/1078-0432.CCR-21-1061. PMID 34315722